CLINICAL TRIAL: NCT06795607
Title: Interventional, Randomized, Single-blind, Placebo-controlled Study to Evaluate the Effect of a Probiotic Formulation Based on SF68® on Body Composition and Low-to-moderate Cardiovascular Risk
Brief Title: Effect of the Probiotic SF68® on Body Composition and Low-to-moderate Cardiovascular Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Francesco Sofi, Associate Professor of Clinical Nutrition, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PrOBesity study
Record Dates: First submitted 2025-01-21; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Probiotic (Experimental): Probiotic food supplement produced by Cerbios-Pharma SA
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): Placebo food supplement
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — The experimental product is a dietary supplement manufactured by Cerbios-Pharma S.A, Each stick contains probiotic live cultures of Enterococcus lactis SF68® at a concentration of 10^9 CFU, phytosterols, 6S-5MeTHF, maltose and silicon dioxide. Study participants will be given N°3 packs each containing 30 stick packs of 1.7 g each, in granulated form in sufficient quantity for the entire duration of the study (12 weeks). Subjects will be required to consume N°1 stick pack of the supplement daily after dinner for 12 continuous weeks. The product should be placed directly on the tongue and should be taken without water. After taking the product, the subject should drink half a glass of water to promote solubilization and transit. The supplement should be stored in a cool, dry place, away from light, moisture and direct heat sources to ensure the viability of the probiotic strain until the expiration date.
  Arms: Probiotic
Dietary Supplement: Placebo — N°1 stick/day of placebo food supplement (i.e., stick without added probiotics), with the same intake modalities as probiotic.
  Arms: Placebo

SUMMARY:
Obesity is a multifactorial disorder of energy balance, characterized by an imbalance between energy intake and energy consumption. In recent decades, the prevalence of obesity has reached epidemic proportions. Advances in scientific research have enabled better characterization of the etiology of obesity, highlighting the potential contribution of factors not traditionally considered to be involved in changes in energy balance and body composition, such as the gut microbiota. Oral administration of probiotics has been proposed as a valid way to modulate the gut ecosystem to promote weight reduction. Preliminary data from a preclinical study in mouse models suggest that the dietary supplement SF68® containing the probiotic Enterococcus lactis as well as phytosterols and (6S)-5-methyltetrahydrofolic acid has the ability to significantly counteract weight gain. In addition to modulating the composition of the gut microbiota, it also has an impact on decreasing the levels of total cholesterol, low-density cholesterol (LDL), triglycerides, homocysteine, IL-1 β and LPS Binding Protein (LBP). Although exercise and diet are the first lines of intervention to be recommended, there are often failures or poor results. There is currently increased interest in alternative and effective shorter-term, non-pharmacological approaches to weight control that involve the use of natural active ingredients. Thus, the aim of this intervention study is to investigate whether a supplementation with SF68® could be beneficial for the weight reduction and the improvement of cardiovascular risk profile of people with overweight or obesity.

ELIGIBILITY:
Inclusion Criteria:

* Obesity (BMI >30 kg/m^2, class I, II, III) and overweight (BMI 25-29.9 kg/ m^2) and concomitant presence of at least one of the following risk factors detected by hematologic examinations performed within 1 year of the baseline screening visit:

  1. Circulating levels of total cholesterol >190 mg/dL, not on drug treatment
  2. Circulating levels of LDL cholesterol >115 mg/dL, not on drug treatment
  3. Circulating levels of triglycerides >150 mg/dL, not on drug treatment
* Ability and willingness to cooperate during the study, adhere to the procedures stipulated in the protocol and comply with its requirements.
* Ability and willingness to complete questionnaires required by the study and to complete all medical examinations required by the protocol.
* Willingness to discontinue the consumption of functional foods and dietary supplements with probiotics, laxatives and body weight control substances starting 15 days before the screening view and until the conclusion of the study.
* Willingness to maintain a healthy and balanced lifestyle for the duration of the study.
* If female subject of childbearing age, must have a negative urine pregnancy test at screening and agree to use a reliable method of contraception throughout the study
* Ability to provide written informed consent.

Exclusion Criteria:

* Use of probiotics continuously, in the two months prior to the start of the study
* Use of other treatments (medications or nutritional programs) that affect body weight or dyslipidemia, gut microbiota, food intake, and/or energy expenditure (e.g., Statins and Fibrates)
* Antibiotic use
* Weight loss or gain > 5 kg in the 3 months prior to the start of the study.
* Pregnant or lactating women and women of childbearing age unwilling to use an adequate contraceptive method and take a pregnancy test at screening.
* Concurrent enrollment in another or similar obesity treatment program

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Waist circumference | 12 weeks
  Changes of waist circumference from baseline assessed through a metric tape

SECONDARY OUTCOMES:
Gut microbiota | 12 weeks
  Changes of gut microbiota from baseline assessed by NGS technology
Short-chain fatty acids (SCFAs) | 12 weeks
  Changes of SCFAs from baseline assessed by gas chromatography
Hemoglobin | 12 weeks
  Changes of hemoglobin from baseline assessed to standard laboratory procedures.
White blood cells | 12 weeks
  Changes of white blood cells from baseline assessed to standard laboratory procedures.
Red blood cells | 12 weeks
  Changes of red blood cells from baseline assessed to standard laboratory procedures.
Platelets | 12 weeks
  Changes of platelets from baseline assessed to standard laboratory procedures.
Glucose | 12 weeks
  Changes of glucose from baseline assessed to standard laboratory procedures.
Insulin | 12 weeks
  Changes of insulin from baseline assessed to standard laboratory procedures.
Glycated hemoglobin | 12 weeks
  Changes of glycated hemoglobin from baseline assessed to standard laboratory procedures.
HOMA index | 12 weeks
  Changes of HOMA index from baseline assessed to standard laboratory procedures.
Total cholesterol | 12 weeks
  Changes of total cholesterol from baseline assessed to standard laboratory procedures.
LDL cholesterol | 12 weeks
  Changes of LDL cholesterol from baseline assessed to standard laboratory procedures.
HDL cholesterol | 12 weeks
  Changes of HDL cholesterol from baseline assessed to standard laboratory procedures.
Triglycerides | 12 weeks
  Changes of triglycerides from baseline assessed to standard laboratory procedures.
AST | 12 weeks
  Changes of AST from baseline assessed to standard laboratory procedures.
ALT | 12 weeks
  Changes of ALT from baseline assessed to standard laboratory procedures.
GGT | 12 weeks
  Changes of GGT from baseline assessed to standard laboratory procedures.
hs-CRP | 12 weeks
  Changes of hs-CRP from baseline assessed to standard laboratory procedures.
Interleukin 1-alpha | 12 weeks
  Changes of interleukin 1-alpha from baseline assessed to standard laboratory procedures.
Interleukin 1-beta | 12 weeks
  Changes of interleukin 1-beta from baseline assessed to standard laboratory procedures.
Interleukin 6 | 12 weeks
  Changes of interleukin 6 from baseline assessed to standard laboratory procedures.
Interleukin 18 | 12 weeks
  Changes of interleukin 18 from baseline assessed to standard laboratory procedures.
Tumor necrosis factor alpha | 12 weeks
  Changes of tumor necrosis factor alpha from baseline assessed to standard laboratory procedures.
Reactive Oxigen Species (ROS) | 12 weeks
  Changes of Reactive Oxigen Species (ROS) from baseline assessed to standard laboratory procedures.
Glutathione | 12 weeks
  Changes of glutathione from baseline assessed to standard laboratory procedures.
Homocysteine | 12 weeks
  Changes of homocysteine from baseline assessed to standard laboratory procedures.
LPS-binding protein | 12 weeks
  Changes of LPS-binding protein from baseline assessed to standard laboratory procedures.
Weight | 12 weeks
  Changes of body weight from baseline assessed through a balance.
Fat mass | 12 weeks
  Changes of fat mass from baseline assessed through a bioelectrical impedance analysis device (Tanita, TBF-410)
Fat-free mass | 12 weeks
  Changes of fat-free mass from baseline assessed through a bioelectrical impedance analysis device (Tanita, TBF-410)
Dietary habits | 12 weeks
  Changes of dietary habits from baseline assessed through the Medi-Lite score, with a total score ranging from 0 to 18, with higher scores meaning a higher adherence to the Mediterranean diet.
Gastrointestinal and systemic symptoms through the GAI score | 12 weeks
  Changes of gastrointestinal and systemic symptoms from baseline assessed through the Global Assessment of Improvement Scale (GAI), with a total score ranging from 0 to 56, with higher scores meaning an improvement of the symptoms
Gastrointestinal and systemic symptoms through the SSS score | 12 weeks
  Changes of gastrointestinal and systemic symptoms from baseline assessed through the Symptom Severity Scale (SSS), with a total score ranging from 0 to 500, with higher scores meaning more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Sofi, Prof., Principal Investigator — Unit of Clinical Nutrition, University Hospital of Careggi Florence, Italy, 50134
Locations (1):
- Careggi University Hospital, Florence, Florence, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borgeraas H, Johnson LK, Skattebu J, Hertel JK, Hjelmesaeth J. Effects of probiotics on body weight, body mass index, fat mass and fat percentage in subjects with overweight or obesity: a systematic review and meta-analysis of randomized controlled trials. Obes Rev. 2018 Feb;19(2):219-232. doi: 10.1111/obr.12626. Epub 2017 Oct 18. PMID 29047207
- [Background] Chung HJ, Yu JG, Lee IA, Liu MJ, Shen YF, Sharma SP, Jamal MA, Yoo JH, Kim HJ, Hong ST. Intestinal removal of free fatty acids from hosts by Lactobacilli for the treatment of obesity. FEBS Open Bio. 2016 Jan 18;6(1):64-76. doi: 10.1002/2211-5463.12024. eCollection 2016 Jan. PMID 27047743
- [Background] Fan Y, Pedersen O. Gut microbiota in human metabolic health and disease. Nat Rev Microbiol. 2021 Jan;19(1):55-71. doi: 10.1038/s41579-020-0433-9. Epub 2020 Sep 4. PMID 32887946
- [Background] Gomes AC, de Sousa RG, Botelho PB, Gomes TL, Prada PO, Mota JF. The additional effects of a probiotic mix on abdominal adiposity and antioxidant Status: A double-blind, randomized trial. Obesity (Silver Spring). 2017 Jan;25(1):30-38. doi: 10.1002/oby.21671. PMID 28008750
- [Background] Holzapfel W, Arini A, Aeschbacher M, Coppolecchia R, Pot B. Enterococcus faecium SF68 as a model for efficacy and safety evaluation of pharmaceutical probiotics. Benef Microbes. 2018 Apr 25;9(3):375-388. doi: 10.3920/BM2017.0148. Epub 2018 Apr 10. PMID 29633645